CLINICAL TRIAL: NCT02605486
Title: Phase I/II Trial of Palbociclib in Combination With Bicalutamide for the Treatment of AR(+) Metastatic Breast Cancer (MBC)
Brief Title: Palbociclib in Combination With Bicalutamide for the Treatment of AR(+) Metastatic Breast Cancer (MBC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-207
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer (MBC)
Keywords: palbociclib; bicalutamide; AR(+); 15-207
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; bicalutamide

ARMS (1):
- Palbociclib in Combination with Bicalutamide (Experimental): This is a non-randomized, open-label, phase I/II trial for patients with AR(+) MBC . There will be a dose finding phase I portion of the study to establish the recommended phase II dose (R2PD). This will be followed by a phase II where efficacy is evaluated. Patients with AR(+)ER(-) breast cancer treated on the phase I at the recommended phase II dose will be counted towards the primary endpoint analysis for the phase II study.
  Interventions: Drug: Palbociclib; Drug: Bicalutamide

INTERVENTIONS:
Drug: Palbociclib
Drug: Bicalutamide

SUMMARY:
The purpose of this study is to test the safety and effectiveness of the investigational drug, palbociclib with bicalutamide for the treatment of triple negative, androgen receptor positive breast cancer.

DETAILED DESCRIPTION:
The study therapy is to be self administered on an outpatient basis. Patients who meet eligibility criteria and sign informed consent to Step 2 may begin treatment on study. Treatment consists of bicalutamide orally once daily and palbociclib will be given orally daily for 3 weeks on followed by 1 week off. A treatment cycle is considered to be 4 weeks. Eligible patients will be evaluated for toxicity every 2 weeks during Cycle #1 and 2, followed by every 4 weeks in subsequent cycles. Toxicity assessment will include history, physical examination including vital signs, and laboratories including complete blood count and comprehensive metabolic panel. Patients will keep a drug diary to document adherence to oral therapy. Radiographic response evaluation per RECIST will occur every 8 weeks (2 cycles) for cycles 1-6 and then every 12 weeks thereafter with high-resolution CT scan. Patients with suspected bone-only lesions must have bone lesions assessed by CT with bone windows or by bone scan at screening.

Phase I: We will use a standard 3+3 design for the dose finding lead in to establish the recommended phase II doses for the combination of palbociclib and bicalutamide. The doses for Phase I will be determined based on the dose level to which the patient is accrued.

Phase II: Treatment consists of bicalutamide orally once daily and palbociclib will be given orally daily for 3 weeks on followed by 1 week off at the doses determined in phase I.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for androgen receptor expression testing (STEP 1) if the following criteria are met:

* Female
* Pathologically confirmed invasive cancer of the breast
* ER/PR status (ER or PR defined as positive if ≥1%; ER/PR is defined as negative if <1%):
* Phase I: Patients may have ER/PR(-) breast cancer.
* HER2 normal (IHC 0-1; FISH < 2.0)
* Non-measurable or measurable, metastatic disease
* Available tissue for AR testing for research purposes

A patient will be eligible for participation in the therapeutic trial (STEP 2) if the following criteria are met:

* Androgen receptor expression testing confirms that the patient's tumor is AR (+). AR is considered positive if ≥1% of cell nuclei are immunoreactive using the Dako antibody (clone AR441). Receptor testing may be performed on either primary tumor specimen or tissue from a metastatic site. Local testing permitted for eligibility but will require confirmation at MSKCC.
* There is no limit to the number of prior chemotherapy or endocrine therapy regimens allowed. Patients with ER(+) AR(+) breast cancer must have had at least 1 prior line of endocrine therapy to be eligible for the phase I portion of the trial.
* At least 2 weeks since last cytotoxic chemotherapy, hormonal therapy, or radiotherapy. Toxicities related to prior therapy must either have returned to grade 1, or baseline (excluding alopecia)
* Patient may receive bisphosphonates/denosumab for the palliation of bone metastases
* If patient has a history of brain metastases or leptomeningeal disease, lesions must be stable for at least 3 months (as documented by either head CT or brain MRI)
* Prior treatment with bicalutamide will not be allowed
* At least 3 weeks from major surgery with full recovery
* ECOG performance status 0-2
* Age 18 years or greater
* Postmenopausal. Use of LHRH agonist permitted.
* Patients must not have another, non-breast, active malignancy that requires treatment.
* The effects of palbociclib on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential must agree to use adequate contraception (barrier method of birth control; abstinence). Women must not breast feed while on study.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow intact palbociclib capsules and bicalutamide tablets.
* Adequate organ and marrow function as defined below (ULN indicates institutional upper limit of normal):

  * Absolute neutrophil count ≥ 1.5 10^9/
  * Hemoglobin ≥ 9.0 g/dL
  * WBC ≥ 3.0 10^9/L
  * Platelets ≥ 100 10^9/L
  * Total bilirubin ≤ 1.5 ULN except for patients with known Gilbert syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 3 institutional ULN
  * Plasma creatinine ≤ 1.5 ULN or Creatinine Clearance > 50 mL/min (calculated by Cockcroft-Gault method)
  * QTc interval ≤ 470 msec

Exclusion Criteria:

* Patients who have not recovered from adverse events of prior therapy to ≤ NCI CTCAEv4.0 Grade 1.
* Patients receiving any other investigational anti-cancer agents.
* Patients who have received prior treatment with a selective CDK4/6 inhibitor
* Patients who have received prior anti-androgen therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib.
* Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (specifically, uncontrolled atrial fibrillation or ventricular dysrhythmias except ventricular premature contractions), or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and women who are breast-feeding.
* Patients with a history of long-QT syndrome or documented family history of long-QT syndrome. Patients who must remain on drugs that prolong the QT interval.
* Palbociclib is a substrate of CYP3A. Caution should be exercised when dosing palbociclib concurrently with CYP3A inducers or inhibitors. Furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
recommended phase II dose (RP2D) (phase I) | 1 year
  We will use a standard 3+3 design for the dose finding lead in to establish the recommended phase II doses for the combination of palbociclib and bicalutamide.
progression free survival (phase II) | 6 monthis
  Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST v 1.1 criteria.

SECONDARY OUTCOMES:
Objective response rate (CR+PR) | 1 year
  Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST v 1.1 criteria.
Clinical benefit rate (CBR) | ≥24 weeks
  (CR+PR+SD)
Progression-free survival | 1 year
  Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST v 1.1 criteria.
Safety and Tolerability by assessing the number of subjects with adverse events | 1 year
  Safety and tolerability will be summarized as per CTCAE version 4 by type and grade, with the maximum grade used as the summary measure per patient across the period of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Gucalp, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/